CLINICAL TRIAL: NCT00083005
Title: A Phase II Trial Combining Estramustine, Docetaxel And Thalidomide In Patients With Androgen-Independent Metastatic Prostate Cancer
Brief Title: Docetaxel, Estramustine, and Thalidomide in Treating Patients With Androgen-Independent Metastatic Adenocarcinoma of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 040132; 04-C-0132; CDR0000361758; NCT00078650 (obsolete NCT alias)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; Thalidomide

INTERVENTIONS:
Drug: docetaxel
Drug: estramustine phosphate sodium
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and estramustine, work in different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of prostate cancer by stopping blood flow to the tumor. Giving chemotherapy together with thalidomide may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel and estramustine together with thalidomide works in treating patients with androgen-independent metastatic adenocarcinoma (cancer) of the prostate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the prostate-specific antigen response in patients with androgen-independent metastatic adenocarcinoma of the prostate treated with docetaxel, estramustine, and thalidomide.

Secondary

* Determine the survival duration in patients treated with this regimen.
* Determine the pharmacokinetics of both docetaxel and thalidomide in patients treated with this regimen.
* Determine whether any pharmacodynamic relationships exist between plasma concentrations of docetaxel and/or thalidomide and clinical activity or toxicity of this regimen in these patients.
* Determine the existence of and quantification of circulating prostate cancer cells in patients before and after treatment with this regimen.
* Determine genotype, with regard to cytochrome P450 2C19 polymorphism, in patients treated with this regimen.
* Correlate genotype with pharmacokinetics and efficacy of this regimen in these patients.
* Determine the changes in molecular markers of angiogenesis (including, but not limited to, serum and urine vascular endothelial growth factor) in patients before and after treatment with this regimen.
* Determine the toxicity profile of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive docetaxel IV over 30 minutes on days 2, 9, and 16, oral thalidomide once daily on days 1-28, and oral estramustine three times daily on days 1-3, 8-10, and 15-17. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 33-60 patients will be accrued for this study within 11-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic disease
  * Androgen-independent disease
* Clinically progressive disease documented by at least 1 of the following parameters:

  * Two consecutively rising prostate-specific antigen (PSA) levels taken at least 1 week apart

    * PSA ≥ 5.0 ng/mL
    * Continued rise in PSA 4 weeks after discontinuation of prior flutamide OR 6 weeks after discontinuation of prior bicalutamide or nilutamide (for patients treated with anti-androgen agents)
  * At least 1 new lesion on bone scan
  * Progressive measurable disease
* Must have undergone bilateral surgical castration OR continue on a gonadotropin-releasing hormone agonist
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count ≥ 100,000/mm^3*
* Hemoglobin ≥ 7.5 g/dL* NOTE: *No transfusions within the past 2 weeks

Hepatic

* AST and ALT < 2.5 times upper limit of normal (ULN)
* Bilirubin < ULN (≤ 3.0 times ULN for patients with Gilbert's syndrome)
* Alkaline phosphatase ≤ 2.5 times ULN OR
* Fractionated hepatic alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* No transient ischemic attacks or cerebrovascular accident within the past 2 years
* No myocardial infarction within the past 6 months
* No uncontrolled congestive heart failure
* No uncontrolled angina pectoris
* No thromboembolic disease

Other

* No peripheral neuropathy ≥ grade 2
* No cognitive impairment that would preclude study participation or giving informed consent
* No other active malignancy within the past 2 years except non-melanoma skin cancer or superficial bladder carcinoma
* Fertile patients must use effective contraception for at least 1 month before, during, and for at least 1 month after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior thalidomide

Chemotherapy

* No prior docetaxel
* No prior estramustine
* No prior chemotherapy for metastatic prostate cancer

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent complementary or alternative therapy that would interact with study drugs
* No concurrent herbal or nutritional products or dietary supplements that would interact with study drugs
* No concurrent aprepitant as secondary prophylaxis or antiemetic treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
PSA response
Toxicity

SECONDARY OUTCOMES:
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Avi S. Retter, MD, Study Chair — Eastchester Center for Cancer Care
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Background] Sissung TM, Danesi R, Kirkland CT, Baum CE, Ockers SB, Stein EV, Venzon D, Price DK, Figg WD. Estrogen receptor alpha and aromatase polymorphisms affect risk, prognosis, and therapeutic outcome in men with castration-resistant prostate cancer treated with docetaxel-based therapy. J Clin Endocrinol Metab. 2011 Feb;96(2):E368-72. doi: 10.1210/jc.2010-2070. Epub 2010 Nov 24. PMID 21106711